CLINICAL TRIAL: NCT00543543
Title: A Randomized, International, Double-Blinded (With In-House Blinding), Controlled With GARDASIL, Dose-Ranging, Tolerability, Immunogenicity, and Efficacy Study of a Multivalent Human Papillomavirus (HPV) L1 Virus-Like Particle (VLP) Vaccine Administered to 16- to 26- Year-Old Women
Brief Title: Broad Spectrum HPV (Human Papillomavirus) Vaccine Study in 16-to 26-Year-Old Women (V503-001)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V503-001; 2007_538
Record Dates: First submitted 2007-10-12; First posted 2007-10-15 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Cervical Cancer; Vulvar Cancer; Vaginal Cancer; Genital Warts; Human Papillomavirus Infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Condylomata Acuminata; Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low-dose V503 (Experimental): V503 (9-Valent Human Papillomavirus [HPV] Vaccine) low-dose 0.5 mL injection in a 3-dose regimen in the base study.
  Interventions: Biological: Experimental: V503
- Mid-dose V503 (Experimental): V503 (9-Valent HPV Vaccine) mid-dose 0.5 mL injection in a 3-dose regimen in the base study. A subset of participants (Cohort 1) received a fourth V503 mid-dose vaccination in the extension study.
  Interventions: Biological: Experimental: V503
- High-dose V503 (Experimental): V503 (9-Valent HPV Vaccine) high-dose 0.5 mL injection in a 3-dose regimen in the base study.
  Interventions: Biological: Experimental: V503
- Gardasil (Active Comparator): Gardasil (4-Valent HPV Vaccine) 0.5 mL injection in a 3-dose regimen in the base study. Participants (Cohort 2) were offered the V503 mid-dose 3-dose regimen in the extension study.
  Interventions: Biological: Comparator: GARDASIL; Biological: Experimental: V503

INTERVENTIONS:
Biological: Comparator: GARDASIL — GARDASIL (quadrivalent HPV [Types 6, 11, 16, and 18] L1 virus-like particle vaccine), 0.5 mL injection in 3 dose regimen
  Arms: Gardasil
Biological: Experimental: V503 — V503 (9-valent HPV [Types 6, 11, 16, 18, 31, 33, 45, 52, and 58] L1 virus-like particle vaccine), 0.5 mL injection in 3 dose regimen (and a fourth injection for Cohort 1 only).

SUMMARY:
The purpose of this study was to evaluate the safety, efficacy, and immunogenicity of V503 in comparison to GARDASIL. The primary hypotheses tested in the study were 1) V503 administered to 16- to 26-year-old adolescents and young women is generally well-tolerated, 2) V503 reduces combined incidence of Human Papillomavirus (HPV) Type 31/33/45/52/58-related disease compared with GARDASIL, and 3) V503 induces non-inferior geometric mean titers for HPV Type 6/11/16/18 antibodies compared with GARDASIL.

DETAILED DESCRIPTION:
The study included a dose-finding evaluation of a 3-dose regimen of V503 and GARDASIL, a safety/efficacy evaluation of a 3-dose regimen of the selected V503 dose formulation and GARDASIL, and an extension consisting of 2 substudies: an evaluation of immune memory in participants receiving a fourth vaccination with V503 (Cohort 1), and an opportunity for participants who received GARDASIL in the Base Study to receive a 3-dose regimen of V503 (Cohort 2).

ELIGIBILITY:
Inclusion Criteria:

* Female between 16- to 26-years-old
* Has never had Pap testing or has only had normal Pap (Papanicolaou) test results
* For the immune memory substudy in the extension (Cohort 1): was randomized to V503 in the base study and was in the per-protocol immunogenicity population for ≥1 HPV type
* For the 3-dose V503 vaccination substudy in the extension (Cohort 2): was randomized to GARDASIL in the base study and received ≥1 dose of GARDASIL

Exclusion Criteria:

* History of an abnormal cervical biopsy result
* History of a positive test for HPV
* History of external genital/vaginal warts
* Currently a user of any illegal drugs or an alcohol abuser
* History of severe allergic reaction that required medical attention
* Are pregnant
* Received marketed HPV vaccine or participated in an HPV trial
* Currently enrolled in a clinical trial
* Currently has or has a history of certain medical conditions or is currently taking or has taken certain medications (details will be discussed at the time of consent.)

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14840 (Actual)
Dates: Start 2007-09-24 (Actual); Primary Completion 2013-04-10 (Actual); Study Completion 2016-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Luxembourg A, Brown D, Bouchard C, Giuliano AR, Iversen OE, Joura EA, Penny ME, Restrepo JA, Romaguera J, Maansson R, Moeller E, Ritter M, Chen J. Phase II studies to select the formulation of a multivalent HPV L1 virus-like particle (VLP) vaccine. Hum Vaccin Immunother. 2015;11(6):1313-22. doi: 10.1080/21645515.2015.1012010. PMID 25912208
- [Result] Joura EA, Giuliano AR, Iversen OE, Bouchard C, Mao C, Mehlsen J, Moreira ED Jr, Ngan Y, Petersen LK, Lazcano-Ponce E, Pitisuttithum P, Restrepo JA, Stuart G, Woelber L, Yang YC, Cuzick J, Garland SM, Huh W, Kjaer SK, Bautista OM, Chan IS, Chen J, Gesser R, Moeller E, Ritter M, Vuocolo S, Luxembourg A; Broad Spectrum HPV Vaccine Study. A 9-valent HPV vaccine against infection and intraepithelial neoplasia in women. N Engl J Med. 2015 Feb 19;372(8):711-23. doi: 10.1056/NEJMoa1405044. PMID 25693011
- [Result] Chen YH, Gesser R, Luxembourg A. A seamless phase IIB/III adaptive outcome trial: design rationale and implementation challenges. Clin Trials. 2015 Feb;12(1):84-90. doi: 10.1177/1740774514552110. Epub 2014 Oct 1. PMID 25278227
- [Result] Luxembourg A, Bautista O, Moeller E, Ritter M, Chen J. Design of a large outcome trial for a multivalent human papillomavirus L1 virus-like particle vaccine. Contemp Clin Trials. 2015 May;42:18-25. doi: 10.1016/j.cct.2015.02.009. Epub 2015 Mar 3. PMID 25749310
- [Result] Pitisuttithum P, Velicer C, Luxembourg A. 9-Valent HPV vaccine for cancers, pre-cancers and genital warts related to HPV. Expert Rev Vaccines. 2015;14(11):1405-19. doi: 10.1586/14760584.2015.1089174. Epub 2015 Sep 14. PMID 26366475
- [Result] Moreira ED Jr, Block SL, Ferris D, Giuliano AR, Iversen OE, Joura EA, Kosalaraksa P, Schilling A, Van Damme P, Bornstein J, Bosch FX, Pils S, Cuzick J, Garland SM, Huh W, Kjaer SK, Qi H, Hyatt D, Martin J, Moeller E, Ritter M, Baudin M, Luxembourg A. Safety Profile of the 9-Valent HPV Vaccine: A Combined Analysis of 7 Phase III Clinical Trials. Pediatrics. 2016 Aug;138(2):e20154387. doi: 10.1542/peds.2015-4387. Epub 2016 Jul 15. PMID 27422279
- [Result] Huh WK, Joura EA, Giuliano AR, Iversen OE, de Andrade RP, Ault KA, Bartholomew D, Cestero RM, Fedrizzi EN, Hirschberg AL, Mayrand MH, Ruiz-Sternberg AM, Stapleton JT, Wiley DJ, Ferenczy A, Kurman R, Ronnett BM, Stoler MH, Cuzick J, Garland SM, Kjaer SK, Bautista OM, Haupt R, Moeller E, Ritter M, Roberts CC, Shields C, Luxembourg A. Final efficacy, immunogenicity, and safety analyses of a nine-valent human papillomavirus vaccine in women aged 16-26 years: a randomised, double-blind trial. Lancet. 2017 Nov 11;390(10108):2143-2159. doi: 10.1016/S0140-6736(17)31821-4. Epub 2017 Sep 5. PMID 28886907
- [Derived] Joura E, Kjaer SK, Bautista O, Luxembourg A, Saah A, Giuliano A. Effect of Prior 9-Valent Human Papillomavirus Vaccination on Subsequent Lower Genital Tract Dysplasia After Cervical Excisional Surgery. Obstet Gynecol. 2026 Jan 1;147(1):73-82. doi: 10.1097/AOG.0000000000006113. Epub 2025 Oct 30. PMID 41166720
- [Derived] Kjaer SK, Nygard M, Sundstrom K, Munk C, Berger S, Dzabic M, Fridrich KE, Waldstrom M, Sorbye SW, Bautista O, Group T, Luxembourg A. Long-term effectiveness of the nine-valent human papillomavirus vaccine in Scandinavian women: interim analysis after 8 years of follow-up. Hum Vaccin Immunother. 2021 Apr 3;17(4):943-949. doi: 10.1080/21645515.2020.1839292. Epub 2020 Dec 16. PMID 33326342
- [Derived] Giuliano AR, Joura EA, Garland SM, Huh WK, Iversen OE, Kjaer SK, Ferenczy A, Kurman RJ, Ronnett BM, Stoler MH, Bautista OM, Moeller E, Ritter M, Shields C, Luxembourg A. Nine-valent HPV vaccine efficacy against related diseases and definitive therapy: comparison with historic placebo population. Gynecol Oncol. 2019 Jul;154(1):110-117. doi: 10.1016/j.ygyno.2019.03.253. Epub 2019 Apr 11. PMID 30982556
- [Derived] Garland SM, Pitisuttithum P, Ngan HYS, Cho CH, Lee CY, Chen CA, Yang YC, Chu TY, Twu NF, Samakoses R, Takeuchi Y, Cheung TH, Kim SC, Huang LM, Kim BG, Kim YT, Kim KH, Song YS, Lalwani S, Kang JH, Sakamoto M, Ryu HS, Bhatla N, Yoshikawa H, Ellison MC, Han SR, Moeller E, Murata S, Ritter M, Sawata M, Shields C, Walia A, Perez G, Luxembourg A. Efficacy, Immunogenicity, and Safety of a 9-Valent Human Papillomavirus Vaccine: Subgroup Analysis of Participants From Asian Countries. J Infect Dis. 2018 Jun 5;218(1):95-108. doi: 10.1093/infdis/jiy133. PMID 29767739
- [Derived] Ruiz-Sternberg AM, Moreira ED Jr, Restrepo JA, Lazcano-Ponce E, Cabello R, Silva A, Andrade R, Revollo F, Uscanga S, Victoria A, Guevara AM, Luna J, Plata M, Dominguez CN, Fedrizzi E, Suarez E, Reina JC, Ellison MC, Moeller E, Ritter M, Shields C, Cashat M, Perez G, Luxembourg A. Efficacy, immunogenicity, and safety of a 9-valent human papillomavirus vaccine in Latin American girls, boys, and young women. Papillomavirus Res. 2018 Jun;5:63-74. doi: 10.1016/j.pvr.2017.12.004. Epub 2017 Dec 19. PMID 29269325
- [Derived] Moreira ED, Giuliano AR, de Hoon J, Iversen OE, Joura EA, Restrepo J, Van Damme P, Vandermeulen C, Ellison MC, Krick A, Shields C, Heiles B, Luxembourg A. Safety profile of the 9-valent human papillomavirus vaccine: assessment in prior quadrivalent HPV vaccine recipients and in men 16 to 26 years of age. Hum Vaccin Immunother. 2018 Feb 1;14(2):396-403. doi: 10.1080/21645515.2017.1403700. Epub 2017 Dec 14. PMID 29211620
- [Derived] Guevara A, Cabello R, Woelber L, Moreira ED Jr, Joura E, Reich O, Shields C, Ellison MC, Joshi A, Luxembourg A. Antibody persistence and evidence of immune memory at 5years following administration of the 9-valent HPV vaccine. Vaccine. 2017 Sep 5;35(37):5050-5057. doi: 10.1016/j.vaccine.2017.07.017. Epub 2017 Aug 5. PMID 28789851
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=V503-001&kw=V503-001&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 15,334 participants were screened and 14,840 were randomized into the study.
Period: Base Study
Arm/Group | Low-dose V503 | Mid-dose V503 | High-dose V503 | Gardasil
Started | 315 | 7106 | 310 | 7109
Completed 3 Vaccinations | 300 | 6928 | 297 | 6934
Completed | 295 (Follow-up was up to 7 months) | 5854 (Follow-up was up to 54 months) | 296 (Follow-up was up to 7 months) | 5887 (Follow-up was up to 54 months)
Not Completed | 20 | 1252 | 14 | 1222
Not completed — Adverse Event | 1 | 11 | 0 | 5
Not completed — Lost to Follow-up | 12 | 749 | 9 | 701
Not completed — Physician Decision | 0 | 4 | 0 | 7
Not completed — Protocol Violation | 0 | 6 | 0 | 6
Not completed — Withdrawal by Subject | 7 | 482 | 5 | 503
Period: Extension Study
Arm/Group | Low-dose V503 | Mid-dose V503 | High-dose V503 | Gardasil
Started | 0 (This group did not participate in the Extension Study) | 150 (Cohort 1) | 0 (This group did not participate in the Extension Study) | 3050 (Cohort 2)
Completed | 0 | 150 | 0 | 2824
Not Completed | 0 | 0 | 0 | 226
Not completed — Adverse Event | 0 | 0 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 77
Not completed — Physician Decision | 0 | 0 | 0 | 7
Not completed — Pregnancy | 0 | 0 | 0 | 6
Not completed — Protocol Violation | 0 | 0 | 0 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 120

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose V503 | Mid-dose V503 | High-dose V503 | Gardasil | Total
Number analyzed (Participants) | 315 | 7106 | 310 | 7109 | 14840
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.7 (2.4) | 21.9 (2.5) | 21.9 (2.4) | 21.8 (2.5) | 21.9 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 315 | 7106 | 310 | 7109 | 14840
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Base Study: Combined Incidence of HPV Type 31/33/45/52/58-related Disease (Test of Hypothesis)
Description: HPV Type 31/33/45/52/58-related high-grade Cervical Intraepithelial Neoplasia (CIN 2/3), Adenocarcinoma in Situ (AIS), Invasive Cervical Carcinoma, high-grade Vulvar Intraepithelial Neoplasia (VIN 2/3), high-grade Vaginal Intraepithelial Neoplasia (VaIN 2/3), vulvar cancer, or vaginal cancer were determined by clinical/pathologic criteria and positive Polymerase Chain Reaction (PCR) assay for virus subtype. This outcome measure reports data based on the protocol-specified plan of conducting hypothesis testing when at least 30 cases had accumulated. The cutoff date for this analysis was 10 April 2013. Disease incidence was defined as the number of primary efficacy cases per 10,000 person-years of follow-up in a treatment arm.
Time Frame: From Day 1 until >=30 cases accumulate, up to Month 54 in the base study
Population: The Per-protocol Efficacy population included all participants who received all 3 vaccinations of mid-dose V503 or Gardasil within acceptable day ranges, were seronegative at Day 1 and PCR negative at Day 1 through Day 7 to the relevant HPV types, and had at least 1 follow-up visit following Month 7.
Measure: Number; unit: Cases per 10,000 person-years follow-up
Arm/Group | Mid-dose V503 | Gardasil
Number analyzed (Participants) | 6016 | 6017
Cases per 10,000 person-years follow-up | 0.5 | 15.8
Statistical Analysis 1: Comparison: Mid-dose V503 vs Gardasil; Test type: Superiority or Other; p < 0.0001, Exact test, 1-sided; Vaccine efficacy = 96.7, 95% CI 2-sided [80.9 to 99.8] — Vaccine efficacy = 100 * [1 - (incidence rate with V503 / incidence rate with Gardasil)]. The pre-specified success criterion was a lower bound of the 95% confidence interval of observed efficacy of >25%

2. Primary Outcome: Base Study: Combined Incidence of HPV Type 31/33/45/52/58-related Disease (End-of-study Update)
Description: HPV Type 31/33/45/52/58-related high-grade Cervical Intraepithelial Neoplasia (CIN 2/3), Adenocarcinoma in Situ (AIS), Invasive Cervical Carcinoma, high-grade Vulvar Intraepithelial Neoplasia (VIN 2/3), high-grade Vaginal Intraepithelial Neoplasia (VaIN 2/3), vulvar cancer, or vaginal cancer were determined by clinical/pathologic criteria and positive Polymerase Chain Reaction (PCR) assay for virus subtype. This outcome measure reports cumulative study data through 10 March 2014. Disease incidence was defined as the number of primary efficacy cases per 10,000 person-years of follow-up in a treatment arm.
Time Frame: Up to Month 54 in the base study
Population: as for outcome 1
Measure: Number; unit: Cases per 10,000 person-years follow-up
Arm/Group | Mid-dose V503 | Gardasil
Number analyzed (Participants) | 6016 | 6017
Cases per 10,000 person-years follow-up | 0.5 | 19.0
Statistical Analysis 1: Comparison: Mid-dose V503 vs Gardasil; Test type: Superiority or Other; Exact test, 1-sided; Vaccine efficacy = 97.4, 95% CI 2-sided [85.0 to 99.9] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Base Study: Geometric Mean Titers (GMTs) to HPV Types 6/11/16/18/31/33/45/52/58
Description: Serum antibodies to HPV types 6/11/16/18/31/33/45/52/58 were measured with a Competitive Luminex Immunoassay. Titers are reported in milli Merck Units/mL. Statistical analysis was performed only for HPV types contained in both vaccines.
Time Frame: 4 weeks postdose 3 in the base study
Population: The Per-protocol Immunogenicity population included all participants who were not protocol violators, received all 3 vaccinations of mid-dose V503 or Gardasil within acceptable ranges, were seronegative at Day 1 and PCR negative from Day 1- Month 7 for the relevant HPV types, and had a Month 7 serum sample collected within an acceptable range
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck U/mL
Arm/Group | Mid-dose V503 | Gardasil
Number analyzed (Participants) | 6792 | 6795
milli Merck U/mL
  Anti-HPV Type 6 (n=3993, 3975) | 893.1 [871.7 to 915.1] | 875.2 [854.2 to 896.8]
  Anti-HPV Type 11 (n=3995, 3982) | 666.3 [649.6 to 683.4] | 830.0 [809.2 to 851.4]
  Anti-HPV Type 16 (n=4032, 4062) | 3131.1 [3057.1 to 3206.9] | 3156.6 [3082.3 to 3232.7]
  Anti-HPV Type 18 (n=4539, 4541) | 804.6 [782.7 to 827.1] | 678.7 [660.2 to 697.7]
  Anti-HPV Type 31 (n=4466, 4377) | 658.4 [636.7 to 680.9] | 9.7 [9.4 to 10.1]
  Anti-HPV Type 33 (n=4702, 4691) | 415.9 [405.6 to 426.4] | NA [NA to NA] — The GMT value was <4 milli Merck U/mL
  Anti-HPV Type 45 (n=4792, 4750) | 252.8 [246.2 to 259.6] | NA [NA to NA] — The GMT value was <3 milli Merck U/mL
  Anti-HPV Type 52 (n=4455, 4335) | 379.7 [371.6 to 388.0] | NA [NA to NA] — The GMT value was <3 milli Merck U/mL
  Anti-HPV Type 58 (n=4486, 4446) | 482.5 [469.9 to 495.3] | NA [NA to NA] — The GMT value was <4 milli Merck U/mL
Statistical Analysis 1: Comparison: Mid-dose V503 vs Gardasil; Anti-HPV Type 6; Test type: Non-Inferiority or Equivalence — Non-inferiority required that the lower bound of the two-sided confidence interval (CI) of the GMT ratio was >0.67; p < 0.001, ANOVA; GMT ratio = 1.02, 95% CI 2-sided [0.99 to 1.06] — GMT ratio = GMT (V503) / GMT (Gardasil)
Statistical Analysis 2: Comparison: Mid-dose V503 vs Gardasil; Anti-HPV Type 11; Test type: Non-Inferiority or Equivalence — Non-inferiority required that the lower bound of the two-sided CI of the GMT ratio was >0.67; p < 0.001, ANOVA; GMT ratio = 0.80, 95% CI 2-sided [0.77 to 0.83] — GMT ratio = GMT (V503) / GMT (Gardasil)
Statistical Analysis 3: Comparison: Mid-dose V503 vs Gardasil; Anti-HPV Type 16; Test type: Non-Inferiority or Equivalence — Non-inferiority required that the lower bound of the two-sided CI of the GMT ratio was >0.67; p < 0.001, ANOVA; GMT ratio = 0.99, 95% CI 2-sided [0.96 to 1.03] — GMT ratio = GMT (V503) / GMT (Gardasil)
Statistical Analysis 4: Comparison: Mid-dose V503 vs Gardasil; Anti-HPV Type 18; Test type: Non-Inferiority or Equivalence — Non-inferiority required that the lower bound of the two-sided CI of the GMT ratio was >0.67; p < 0.001, ANOVA; GMT ratio = 1.19, 95% CI 2-sided [1.14 to 1.23] — GMT ratio = GMT (V503) / GMT (Gardasil)

4. Other Pre Specified Outcome: Extension Study: Geometric Mean Titers to HPV Types 6/11/16/18/31/33/45/52/58 at Predose 4
Description: Serum antibodies to HPV types 6/11/16/18/31/33/45/52/58 were measured with a Competitive Luminex Immunoassay. Titers are reported in milli Merck Units/mL. This outcome measure applied to Cohort 1 participants only.
Time Frame: Month 60: predose 4 in the Extension Study (Cohort 1)
Population: All participants in Cohort 1 who received all 3 vaccinations of mid-dose V503 in the Base Study, were seronegative at Day 1 and PCR negative from Day 1 to Month 7 for the relevant HPV types, had no other violation that could interfere with evaluation of immune response, and provided post-dose 4 serum.
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck U/mL
Groups:
- Extension Study: Mid-dose V503 (Cohort 1): V503 mid-dose 0.5 mL injection in a 3-dose regimen in the Base Study. A subset of participants (Cohort 1) received a fourth V503 mid-dose vaccination in the extension study.
Arm/Group | Extension Study: Mid-dose V503 (Cohort 1)
Number analyzed (Participants) | 150
milli Merck U/mL
  Anti-HPV Type 6 (n=101) | 143.1 [117.9 to 173.7]
  Anti-HPV Type 11 (n=112) | 82.9 [68.1 to 100.9]
  Anti-HPV Type 16 (n=128) | 324.4 [266.7 to 394.7]
  Anti-HPV Type 18 (n=142) | 62.5 [49.5 to 78.9]
  Anti-HPV Type 31 (n=135) | 69.2 [56.6 to 84.4]
  Anti-HPV Type 33 (n=141) | 44.7 [37.0 to 54.1]
  Anti-HPV Type 45 (n=148) | 20.8 [17.0 to 25.5]
  Anti-HPV Type 52 (n=134) | 33.7 [27.6 to 41.1]
  Anti-HPV Type 58 (n=132) | 50.9 [40.9 to 63.3]

5. Primary Outcome: Base Study: Percentage of Participants With One or More Adverse Event
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE.
Time Frame: Up to Month 7 (low- and high-dose V503) or up to Month 54 (mid-dose V503 and Gardasil)
Population: The analysis population included all participants who received >=1 vaccination and had safety follow-up
Measure: Number; unit: Percentage of participants
Groups:
- Low-dose V503: V503 (9-Valent HPV Vaccine) low-dose 0.5 mL injection in a 3-dose regimen in the base study.
Arm/Group | Low-dose V503 | Mid-dose V503 | High-dose V503 | Gardasil
Number analyzed (Participants) | 310 | 7071 | 305 | 7078
Percentage of participants | 92.6 | 94.2 | 92.8 | 91.1

6. Primary Outcome: Base Study: Percentage of Participants With One or More Injection-site Adverse Event
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. AEs such as redness, swelling, and pain/tenderness/soreness at the injection site were recorded.
Time Frame: Up to Day 5 after any vaccination
Population: The analysis population included all participants who received >=1 vaccination and had safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | Low-dose V503 | Mid-dose V503 | High-dose V503 | Gardasil
Number analyzed (Participants) | 310 | 7071 | 305 | 7078
Percentage of participants | 87.7 | 90.7 | 90.5 | 84.9

7. Primary Outcome: Base Study: Percentage of Participants With One or More Non-injection-site (Systemic) Adverse Event
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. Systemic AEs were those not categorized as injection-site AEs.
Time Frame: Up to Day 15 after any vaccination
Population: The analysis population included all participants who received >=1 vaccination and had safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | Low-dose V503 | Mid-dose V503 | High-dose V503 | Gardasil
Number analyzed (Participants) | 310 | 7071 | 305 | 7078
Percentage of participants | 53.5 | 55.8 | 51.1 | 54.9

8. Primary Outcome: Base Study: Percentage of Participants With One or More Vaccine-related Adverse Event
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. An AE that is judged by the investigator to be "definitely related," "probably related," or "possibly related" to the study drug is defined as a vaccine-related AE.
Time Frame: Up to Month 7 (low- and high-dose V503) or up to Month 54 (mid-dose V503 and Gardasil)
Population: The analysis population included all participants who received >=1 vaccination and had safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | Low-dose V503 | Mid-dose V503 | High-dose V503 | Gardasil
Number analyzed (Participants) | 310 | 7071 | 305 | 7078
Percentage of participants | 90.0 | 92.2 | 92.8 | 87.6

9. Primary Outcome: Base Study: Percentage of Participants With Study Medication Withdrawn Due to an Adverse Event
Description: An adverse event is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an adverse event.
Time Frame: Up to Month 6
Population: The analysis population included all participants who received >=1 vaccination and had safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | Low-dose V503 | Mid-dose V503 | High-dose V503 | Gardasil
Number analyzed (Participants) | 310 | 7071 | 305 | 7078
Percentage of participants | 0.6 | 0.1 | 0.0 | 0.1

10. Secondary Outcome: Base Study: Combined Incidence of HPV Type 31/33/45/52/58-related Persistent Infection
Description: Combined Incidence of HPV Type 31/33/45/52/58-related persistent infection as determined by clinical/pathologic criteria and positive Polymerase Chain Reaction (PCR) assay for virus subtype. Persistent infection was defined as infection detected in samples from >=2 consecutive visits 6 months (+/-1 month visit window) or longer apart. Incidence was defined as the number of cases of persistent infection per 10,000 person-years of follow-up in a treatment arm.
Time Frame: Up to Month 54 in the base study
Population: as for outcome 1
Measure: Number; unit: Cases per 10,000 person-years follow-up
Arm/Group | Mid-dose V503 | Gardasil
Number analyzed (Participants) | 5941 | 5955
Cases per 10,000 person-years follow-up | 21.5 | 538.8
Statistical Analysis 1: Comparison: Mid-dose V503 vs Gardasil; Test type: Superiority or Other; Vaccine efficacy = 96.0, 95% CI 2-sided [94.6 to 97.1] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Base Study: Percentage of Participants Who Are Seropositive for HPV Types 6/11/16/18/31/33/45/52/58
Description: Serum antibodies to HPV types were measured with a Competitive Luminex Immunoassay. The serostatus cutoffs (milli Merck U/mL) for HPV types were as follows: HPV Type 6: ≥30; HPV Type 11: ≥16; HPV Type 16: ≥20; HPV Type 18: ≥24; HPV Type 31: ≥10; HPV Types 33, 45, 52, and 58: ≥8.
Time Frame: 4 weeks postdose 3
Population: The Per-protocol Immunogenicity population included all participants who were not protocol violators, received all 3 vaccinations of mid-dose V503 or Gardasil within acceptable ranges, were seronegative at Day 1 and PCR negative from Day 1 - Month 7 for the relevant HPV types, and had a Month 7 serum sample collected within an acceptable range
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Mid-dose V503 | Gardasil
Number analyzed (Participants) | 6792 | 6795
Percentage of participants
  Anti-HPV Type 6 (n=3993, 3975) | 99.8 [99.6 to 99.9] | 99.8 [99.7 to 99.9]
  Anti-HPV Type 11 (n=3995, 3982) | 100 [99.9 to 100] | 99.9 [99.8 to 100]
  Anti-HPV Type 16 (n=4032, 4062) | 100 [99.9 to 100] | 100 [99.8 to 100]
  Anti-HPV Type 18 (n=4539, 4541) | 99.8 [99.7 to 99.9] | 99.7 [99.5 to 99.8]
  Anti-HPV Type 31 (n=4466, 4377) | 99.8 [99.6 to 99.9] | 50.1 [48.7 to 51.6]
  Anti-HPV Type 33 (n=4702, 4691) | 99.7 [99.5 to 99.9] | 12.7 [11.8 to 13.7]
  Anti-HPV Type 45 (n=4792, 4750) | 99.6 [99.4 to 99.8] | 9.2 [8.4 to 10.0]
  Anti-HPV Type 52 (n=4455, 4335) | 99.8 [99.6 to 99.9] | 2.6 [2.2 to 3.1]
  Anti-HPV Type 58 (n=4486, 4446) | 99.8 [99.6 to 99.9] | 20.4 [19.2 to 21.6]

12. Other Pre Specified Outcome: Extension Study: Geometric Mean Titers to HPV Types 6/11/16/18/31/33/45/52/58 at Day 7 Postdose 4
Description: as for outcome 4
Time Frame: Month 60 + 1 week: Day 7 postdose 4 in the Extension Study (Cohort 1)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck U/mL
Arm/Group | Extension Study: Mid-dose V503 (Cohort 1)
Number analyzed (Participants) | 150
milli Merck U/mL
  Anti-HPV Type 6 (n=109) | 2180.5 [1826.2 to 2603.7]
  Anti-HPV Type 11 (n=109) | 2228.7 [1852.5 to 2681.3]
  Anti-HPV Type 16 (n=126) | 7986.3 [6795.7 to 9385.6]
  Anti-HPV Type 18 (n=138) | 2399.0 [2049.4 to 2808.1]
  Anti-HPV Type 31 (n=131) | 1462.2 [1263.9 to 1691.5]
  Anti-HPV Type 33 (n=137) | 1709.0 [1466.7 to 1991.2]
  Anti-HPV Type 45 (n=144) | 323.0 [277.2 to 376.5]
  Anti-HPV Type 52 (n=131) | 1078.1 [907.2 to 1281.2]
  Anti-HPV Type 58 (n=129) | 1801.8 [1530.5 to 2121.2]

13. Other Pre Specified Outcome: Extension Study: Geometric Mean Titers to HPV Types 6/11/16/18/31/33/45/52/58 at Day 28 Postdose 4
Description: as for outcome 4
Time Frame: Month 61: 28 days postdose 4 in the Extension Study (Cohort 1)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck U/mL
Arm/Group | Extension Study: Mid-dose V503 (Cohort 1)
Number analyzed (Participants) | 150
milli Merck U/mL
  Anti-HPV Type 6 (n=109) | 2585.0 [2239.5 to 2983.8]
  Anti-HPV Type 11 (n=109) | 2548.7 [2191.4 to 2964.3]
  Anti-HPV Type 16 (n=123) | 10904.3 [9605.6 to 12378.7]
  Anti-HPV Type 18 (n=137) | 2907.9 [2531.1 to 3340.7]
  Anti-HPV Type 31 (n=130) | 1745.4 [1538.8 to 1979.8]
  Anti-HPV Type 33 (n=136) | 2094.9 [1848.7 to 2373.9]
  Anti-HPV Type 45 (n=143) | 440.0 [386.9 to 500.4]
  Anti-HPV Type 52 (n=129) | 1131.5 [991.6 to 1291.1]
  Anti-HPV Type 58 (n=127) | 2024.6 [1803.1 to 2273.2]

ADVERSE EVENTS:
Time Frame: Base Study: SAEs up to Month (M) 7 (low- and high-dose V503) or up to M54 (mid-dose V503 and Gardasil); non-serious AEs up to Day 15 after vaccination. Cohort 1: SAEs M60 to 61; non-serious AEs up to Day 15 after vaccination 4. Cohort 2: SAEs M60 to 67.
Description: The analysis population included all participants who received >=1 vaccination and had safety follow-up. Non-serious AEs were not solicited in Extension Cohort 2; however, some non-serious AEs were voluntarily reported.
Groups:
- Base Study: Low-Dose V503: V503 (9-Valent HPV Vaccine) low-dose 0.5 mL injection in a 3-dose regimen in the base study.
- Base Study: Mid-dose V503: V503 (9-Valent HPV Vaccine) mid-dose 0.5 mL injection in a 3-dose regimen in the base study. A subset of participants (Cohort 1) will receive a fourth V503 mid-dose vaccination in the extension study.
- Base Study: High-dose V503: V503 (9-Valent HPV Vaccine) high-dose 0.5 mL injection in a 3-dose regimen in the base study.
- Base Study: Gardasil: Gardasil (4-Valent HPV Vaccine) 0.5 mL injection in a 3-dose regimen in the base study. Participants (Cohort 2) will be offered the V503 mid-dose 3-dose regimen in the extension study.
- Extension Study: Mid-dose V503 (Cohort 1): V503 (9-Valent HPV Vaccine) mid-dose 0.5 mL fourth dose administration in Base Study participants who were randomized to receive a 3-dose regimen of V503 (9-Valent HPV) mid-dose 0.5 mL (Cohort 1).
- Extension Study: Mid-dose V503 (Cohort 2): V503 (9-Valent HPV Vaccine) mid-dose 0.5 mL 3-dose regimen administration on Base Study participants who were randomized to receive a 3-dose regimen of Gardasil (4-Valent HPV Vaccine) (Cohort 2).
Arm/Group | Base Study: Low-Dose V503 | Base Study: Mid-dose V503 | Base Study: High-dose V503 | Base Study: Gardasil | Extension Study: Mid-dose V503 (Cohort 1) | Extension Study: Mid-dose V503 (Cohort 2)
Serious Adverse Events (participants affected / at risk) | 4/310 | 233/7071 | 5/305 | 184/7078 | 1/150 | 25/3049
Other Adverse Events (participants affected / at risk) | 278/310 | 6551/7071 | 280/305 | 6268/7078 | 130/150 | 89/3049
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study: Low-Dose V503 (N=310) | Base Study: Mid-dose V503 (N=7071) | Base Study: High-dose V503 (N=305) | Base Study: Gardasil (N=7078) | Extension Study: Mid-dose V503 (Cohort 1) (N=150) | Extension Study: Mid-dose V503 (Cohort 2) (N=3049)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cleft lip and palate (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis Meckel's (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Omental infarction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Allergy to vaccine (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 9 (9) | 0 (0) | 16 (16) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post abortion infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukaemic infiltration brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign intracranial hypertension (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial venous sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 36 (38) | 1 (1) | 26 (28) | 0 (0) | 8 (8)
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 4 (4) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Cervix dystocia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
False labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foetal malposition (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Labour complication (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia and bulimia syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia nervosa (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bartholinitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 5 (5) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fallopian tube cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 73 (76) | 2 (2) | 53 (53) | 0 (0) | 3 (3)
Axillary vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholestasis of pregnancy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study: Low-Dose V503 (N=310) | Base Study: Mid-dose V503 (N=7071) | Base Study: High-dose V503 (N=305) | Base Study: Gardasil (N=7078) | Extension Study: Mid-dose V503 (Cohort 1) (N=150) | Extension Study: Mid-dose V503 (Cohort 2) (N=3049)
Nausea (Gastrointestinal disorders) | 22 (23) | 513 (617) | 18 (20) | 459 (551) | 2 (2) | 4 (4)
Injection site erythema (General disorders) | 100 (157) | 2411 (3597) | 91 (140) | 1810 (2564) | 33 (34) | 9 (9)
Injection site pain (General disorders) | 267 (684) | 6360 (15383) | 273 (672) | 5911 (13001) | 124 (128) | 59 (94)
Injection site pruritus (General disorders) | 18 (21) | 389 (494) | 14 (16) | 282 (341) | 1 (1) | 1 (1)
Injection site swelling (General disorders) | 100 (154) | 2836 (4527) | 103 (168) | 2035 (2988) | 49 (51) | 12 (12)
Pyrexia (General disorders) | 30 (35) | 469 (563) | 17 (19) | 463 (550) | 6 (6) | 7 (7)
Influenza (Infections and infestations) | 20 (22) | 312 (343) | 12 (12) | 296 (314) | 4 (5) | 5 (5)
Nasopharyngitis (Infections and infestations) | 10 (11) | 376 (412) | 12 (13) | 389 (420) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 17 (20) | 346 (405) | 11 (13) | 307 (368) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 65 (100) | 1879 (3071) | 66 (106) | 1756 (2788) | 32 (41) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.